CLINICAL TRIAL: NCT04642872
Title: Effects of Infant Constraint Induced Movement Therapy and Infant Bimanual Intensive Therapy in Unilateral Cerebral Palsy. A Randomized Controlled Trial.
Brief Title: Upper Limb Intensive Therapies in Babies With Unilateral Cerebral Palsy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CEU San Pablo University (Other)
Responsible Party: Principal Investigator, Rocio Palomo Carrión, Director, CEU San Pablo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: infant CIMT/BIT
Record Dates: First submitted 2020-11-03; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Infantile Hemiplegia; Upper Extremity Paresis; Family; Constraint Induced Movement Therapy; Bimanual Intensive Therapy
MeSH Terms: conditions — Hemiplegia; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- infant cimt (Experimental)
  Interventions: Other: Infant BIT; Other: Infant CIMT/BIT; Other: Conventional therapy
- Infant BIT (Active Comparator)
  Interventions: Other: Infant CIMT/BIT; Other: Conventional therapy; Other: infant cimt
- Infant CIMT/BIT (Active Comparator)
  Interventions: Other: Infant BIT; Other: Conventional therapy; Other: infant cimt
- Conventional Therapy (Active Comparator)
  Interventions: Other: Infant BIT; Other: Infant CIMT/BIT; Other: infant cimt

INTERVENTIONS:
Other: Infant BIT — Not use of unaffected hand containment. Both hand are use to improve the bimanual coordination
  Arms: Conventional Therapy; Infant CIMT/BIT; infant cimt
Other: Infant CIMT/BIT — Use unaffected hand containment in part of the intervention and then, both hands in bimanual activities without containment.
  Arms: Conventional Therapy; Infant BIT; infant cimt
Other: Conventional therapy — Following the usual therapy in the baby.
  Arms: Infant BIT; Infant CIMT/BIT; infant cimt
Other: infant cimt — use of unaffected hand containment to improve the use of affected hand with unimanual activities
  Arms: Conventional Therapy; Infant BIT; Infant CIMT/BIT

SUMMARY:
mCIMT and BIT are therapies applied in children with hemiplegia which have a great evidence, but not in a early age. This research has the objective to know the effects of this therapies in infants diagnosed of infantile hemiplegia from 9 to 18 months applying 50 hours of dose for both interventions during 10 weeks, executing them at home by familes.

ELIGIBILITY:
Inclusion Criteria:

* Infantile hemiplegia
* Age from 9 months to 18 months.
* No use of the affected upper limb

Exclusion Criteria:

* Associated pathologies
* Epilepsy no controlled with medicins
* No collaborated families

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-07-28 (Actual); Primary Completion 2021-01-18 (Estimated); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
mini Assisting Hand Assesment | 10 weeks
  Bimanual functional performance Assessment in children with hemiplegia from 8 to 18 months.

SECONDARY OUTCOMES:
Satisfaction questionnaire for familes | 10 weeks
  Descriptive questionnaire to obtain the adherence and satisfaction from families in this therapies.

CONTACTS AND LOCATIONS:
Locations (1):
- Hemiweb, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palomo-Carrion R, Pinero-Pinto E, Romay-Barrero H, Escobio-Prieto I, Lillo-Navarro C, Romero-Galisteo RP. Shall we start? Ready, set, go! Toward early intervention in infants with unilateral cerebral palsy. A randomized clinical trial protocol. Ther Adv Chronic Dis. 2022 Nov 14;13:20406223221136059. doi: 10.1177/20406223221136059. eCollection 2022. PMID 36420043